CLINICAL TRIAL: NCT03165149
Title: Effect of a Topical Ketamine on Acute and Chronic Post-mastectomy Pain, Dose Finding - Clinical Study
Brief Title: Effect of a Topical Ketamine on Acute and Chronic Pain, Dose Finding
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Fatma Adel El sherif,MD, lecturer of anesthesia, ICU and pain releif, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 17100205
Record Dates: First submitted 2017-05-23; First posted 2017-05-24 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-10

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Population Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Group (A) (Active Comparator): patients will receive 1mg / kg of Ketamine diluted by 20 ml saline (0.9 % )
  Interventions: Drug: group (A)
- Group (B) (Active Comparator): patients will receive 2 mg /kg of Ketamine diluted by 20 ml saline (0.9 %) a
  Interventions: Drug: group (B)
- Group (C) (Active Comparator): patients will receive 3 mg / kg of Ketamine diluted by 20 ml saline (0.9 %)
  Interventions: Drug: group (c)

INTERVENTIONS:
Drug: group (A) — patients will receive 1mg / kg of Ketamine diluted by 20 ml saline (0.9 % ) and irrigated onto surgical field after hemostats and before skin closure.
  Arms: Group (A)
Drug: group (B) — patients will receive 2 mg /kg of Ketamine diluted by 20 ml saline (0.9 %) and irrigated onto surgical field after hemostasis and before skin closure.
  Arms: Group (B)
Drug: group (c) — patients will receive 3 mg /kg of Ketamine diluted by 20 ml saline (0.9 %) and irrigated onto surgical field after hemostasis and before skin closure.
  Arms: Group (C)

SUMMARY:
The aim of this study is to investigate the effect of addition of different doses of Ketamine locally in acute and chronic post-mastectomy pain after breast cancer surgery and on the probability of developing chronic post-mastectomy pain.

ELIGIBILITY:
Inclusion Criteria:

- American society of heart association class I-II female patients

* aged 18-60 years
* scheduled for modified radical mastectomy with axillary dissection for breast carcinoma

Exclusion Criteria:

* known allergy to the study drugs
* significant cardiac-
* respiratory-
* renal or hepatic disease

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 90 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
the total amount of morphine consumption | 48 hours
  total amount of rescue analgesia

SECONDARY OUTCOMES:
pain intensity | 48 hours
  pain intensity measured by Visual analogue scale

CONTACTS AND LOCATIONS:
Locations (1):
- South Egypt Cancer Instuite, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No